CLINICAL TRIAL: NCT06794918
Title: Investigation of the Effects of Relaxation Exercises Applied to Patients With Type 2 Diabetes on Neuropathic Pain, Fatigue and Sleep Quality
Brief Title: Investigation of the Effects of Relaxation Exercises on Neuropathic Pain, Fatigue and Sleep Quality
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Eren KILIC, lecturer, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ErenKILIC
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Type 2 Diabetes; Progressive Relaxation Exercise; Neuropathic Pain; Fatigue; Sleep Quality
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Neuralgia; Fatigue; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Progressive relaxation exercises will be applied to the experimental group.
  Interventions: Diagnostic Test: progressive relaxation exercise
- no intervention group (No Intervention): The control group will not receive any intervention.

INTERVENTIONS:
Diagnostic Test: progressive relaxation exercise — Researchers will teach individuals pge exercises to help them relax
  Arms: intervention group

SUMMARY:
Relaxation exercises are an important factor in improving diabetes management and quality of life. Diet, exercise, medication and insulin therapy are important components of diabetes management. Among the goals that relaxation exercises should achieve is not only to provide information but also to ensure the patient's active participation in treatment by improving their application skills. Progressive Relaxation Exercises (PGE) are among the effective improvement techniques in the care process. Type 2 diabetes is a common metabolic disease and its chronic complications include neuropathic pain, fatigue and sleep disorders. Nurses play an important role in the care of these patients and the management of such symptoms is at the center of nursing practice. As a result, examining the effects of relaxation exercises on neuropathic pain, fatigue and sleep quality for patients with type 2 diabetes can increase the effectiveness of non-pharmacological approaches in nursing care and improve the quality of life of patients. Such studies have the potential to increase the quality of care and patient satisfaction by supporting the evidence-based practices of nurses. Hypotheses of the Study Hypothesis (H0): Progressive relaxation exercise has no effect on neuropathic pain, fatigue, and sleep quality of individuals with Type 2 diabetes.

Hypothesis (H1): Progressive relaxation exercise has an effect on the neuropathic pain level of individuals with Type 2 diabetes.

Hypothesis (H2): Progressive relaxation exercise has an effect on the fatigue level of individuals with Type 2 diabetes.

Hypothesis (H3): Progressive relaxation exercise has an effect on the sleep quality of individuals with Type 2 diabetes. In light of all this information, the proposed study aimed to investigate the effects of relaxation exercises applied to study groups formed with diabetic patients on neuropathic pain, sleep quality and fatigue.

DETAILED DESCRIPTION:
Research Phases Preliminary Preparation

A comprehensive literature review was conducted to examine the content and structure of previously published studies. Based on this review, the most suitable materials for the purpose of the present study were identified. Among these, the Progressive Relaxation Exercise Audio CD prepared by the Turkish Psychological Association was selected, and the necessary permissions were obtained for its inclusion in the research. Prior to data collection, official approval was obtained from both the hospital administration and the responsible physician of the Endocrinology Inpatient Unit at Erzurum Atatürk Training and Research Hospital.

Progressive Muscle Relaxation

Progressive Muscle Relaxation (PMR) is a self-administered relaxation technique that involves the sequential tensing and releasing of sixteen major muscle groups in the body. During the exercise, deep breathing accompanies the commands to contract and relax each muscle group - muscles are tensed while inhaling and relaxed while exhaling. This method has been recognized as an effective intervention for reducing pain, anxiety, and depression. Additionally, incorporating mindful awareness of breathing has been shown to accelerate the relaxation response.

The steps of the Progressive Muscle Relaxation exercise are as follows:

Step 1: Begin with slow, deep, and rhythmic diaphragmatic breathing through the nose and out through the mouth. The abdomen should remain relaxed, and hands are placed on the lower abdomen to monitor diaphragmatic movement. The abdomen rises during inhalation and falls during exhalation. Chest movement should be minimized, as it may indicate insufficient diaphragmatic engagement.

Step 2: Breathing exercises start with exhalation lasting approximately twice as long as inhalation, a strategy known to promote general relaxation. After exhalation, a brief rest is taken before the next inhalation. Once slow and deep breathing has been repeated several times, participants proceed to the progressive muscle relaxation exercises.

Step 3: During PMR, the major muscle groups - including the feet, legs, hips, abdomen, chest, back, hands, arms, neck, shoulders, and facial muscles - are sequentially tensed while inhaling and relaxed while exhaling. After each muscle group, several deep diaphragmatic breaths are taken to allow short rest periods. At the end of the exercise, all muscle groups are tensed and relaxed simultaneously, and the session concludes with slow, deep breathing.

Implementation of the Study

Patients who met the inclusion criteria in the experimental group performed the Progressive Relaxation Exercises using the Progressive Relaxation Exercise CD in a calm environment, either in a seated or semi-seated comfortable position. The sessions were conducted in designated rooms within the Atatürk University Training and Research Hospital or in alternative suitable settings based on patient preference (such as their homes or nearby family health centers).

The exercises were supervised by the researcher twice a week, while on the remaining days participants performed the exercises independently by listening to the CD for 30 minutes daily over a period of six weeks. The duration and frequency of the sessions were determined by reviewing similar studies in the literature, which generally applied PMR once daily for 30-minute sessions over 6-8 weeks to address fatigue and sleep problems. Considering that the FACIT Fatigue Scale assesses fatigue over the past week and the Pittsburgh Sleep Quality Index (PSQI) assesses sleep quality over the past four weeks, as well as the time required for participants to adapt to relaxation techniques, the six-week daily practice was deemed appropriate. No intervention was administered to the control group during this period.

Procedures Applied to the Experimental Group

Before initiating the intervention, nurses, physicians, and other healthcare personnel working in the Endocrinology Inpatient Unit of Erzurum Atatürk Training and Research Hospital were informed about the study.

All interviews and sessions were conducted in quiet, clean, and well-ventilated education rooms within the Endocrinology Unit or in nearby family health centers where participants could feel comfortable and safe. Depending on availability, participants were grouped into sessions of 2-5 individuals. In the initial session, participants received education on the concept, importance, purpose, benefits, and key considerations of relaxation. Correct breathing techniques - the first step of the relaxation process - were demonstrated and practiced.

Subsequently, participants were taught the definition, importance, and methods of performing Progressive Relaxation Exercises through demonstration and guided practice. Each participant was instructed individually by the researcher to ensure correct technique. The "Relaxation Exercise Audio Recordings" prepared by the Turkish Psychological Association were used as nursing intervention material.

The CD consists of three parts:

The first part explains the purpose of deep relaxation in a 10-minute session.

The second part provides a 30-minute guided relaxation exercise accompanied by water sounds and verbal instructions.

The third part includes 30 minutes of relaxation music only.

In this study, the second part of the CD was used. Before starting the exercise, participants were seated comfortably in a chair and informed that, at home, they could perform the exercise lying on a bed. Following the audio instructions, participants were guided to tense each muscle group while counting to five and then relax, inhaling deeply during tension and exhaling slowly during relaxation. This process was applied to the hands, arms, neck, shoulders, chest, abdomen, hips, legs, feet, and facial muscles - sequentially from the hands to the feet - allowing full-body relaxation.

To enhance comfort and effectiveness, participants were advised to wear loose clothing and perform the exercises in a quiet setting. Each educational session lasted 30 minutes.

The exercises were performed twice weekly under supervision and daily at home for six weeks using the provided audio materials. Participants received instructions on how and when to practice at home and were shown how to use the recordings. They were also provided with the researcher's phone number for consultation when needed. A WhatsApp group was created to monitor adherence, with weekly phone calls and reminder messages sent to participants throughout the six-week period to encourage daily practice compliance.

This research was planned as a randomized controlled experimental study. The research will be conducted with Type 2 DM patients who apply to Erzurum Ataturk Education and Research Hospital Endocrinology Polyclinic/Inpatient Service. The universe of the research will consist of patients who apply to Erzurum Ataturk Education and Research Hospital Endocrinology Polyclinic/Inpatient Service and are followed up and diagnosed with Type 2 DM. The sample size of the research was calculated using the G*Power 3.1. 9.6 program. In the calculation, the 2-group (Experimental Group, Control Group) and 2-measurement (Pretest, Posttest) research design was taken into consideration and the sample calculation was made for the independent groups t-test. In the calculation, medium effect size (d = 0.50), 5% margin of error (α = 0.05) and 80% power (1-β = 0.80) were taken into account, and the sample number for each group was calculated as 40. Considering the possibility of data loss, the sample size for each group was increased by 10% and it was planned to include 44 people in each group, a total of 88 people in the sample. In collecting the research data; the Patient Identification Form prepared by the researcher with literature including the socio-demographic and disease-related characteristics of the patients and the patient's metabolic values, the S-LANSS Neuropathic Pain Scale to assess the neuropathic pain levels of diabetic individuals, the FACIT-Fatigue Scale to assess the fatigue levels of diabetic individuals and the Pittsburgh Sleep Quality Index (PUKI) Scale to assess the sleep quality of diabetic patients will be used. The research data will be analyzed using the SPSS 26.0 (Statistical Package for the Social Sciences) program. Frequency, percentage, mean and standard deviation values will be calculated in the evaluation of descriptive data. The significance level will be accepted as 0.05 (p < 0.05) in the analyses. The Shapiro Wilks test will be used for normal distribution. The mean scores of the scales used to evaluate neuropathic pain, fatigue, and sleep quality of the experimental and control groups will be compared between the groups using a t-test in independent groups, and the comparison of the mean pre-test and post-test scores within the group will be evaluated using a t-test in dependent groups.

ELIGIBILITY:
Inclusion Criteria for the Study

* Those diagnosed with Type II DM for at least six months,
* Those aged between 18 and 65,
* Those who are literate,
* Those taking insulin and oral antidiabetic treatment,
* Those without a psychiatric illness,
* Those without any communication problems (vision, hearing, or speech),
* Those not using sleeping pills,
* Those with a Pittsburgh Sleep Quality Index average score of 5 or higher,
* Those with an S-LANSS average score of 12 or higher,
* Those with a FACIT (Fatigue Scale) average score of less than 30. 3.9. Exclusion Criteria for the Study
* Those with a diabetic foot wound,
* Those with an amputation,
* Those with a malignant disease,
* Those with COPD or asthma,
* Those who discontinued the Progressive Relaxation Exercise program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2026-02-07 (Estimated)

PRIMARY OUTCOMES:
S-LANSS Neuropathic Pain Scale | 6 weeks
  The S-LANSS pain score is based on the patient's assessment of the worst pain they have felt in the past week. This scale consists of a total of 7 questions; the first 5 questions are about pain symptoms, while the last 2 questions are aimed at determining the presence of allodynia (pain in response to a stimulus that is normally painless) and decreased pain sensation. The questions are answered only with "yes" or "no". Patients can receive a score between 0 and 24 on the test. The test results of patients who score 12 or higher support neuropathic pain, while the results of patients who score below 12 indicate non-neuropathic pain. (Bennett et al., 2005; Weingarten et al., 2007) The validity and reliability study of the S-LANSS Neuropathic Pain Scale was conducted in 2008 by Dr. Emine Rabia KOÇ. The reliability coefficients (Cronbach alpha value) between the items in the 1st and 2nd applications of the S-LANSS pain score were calculated as 0.74. The correlation coefficients for each
FACIT- (Fatigue) Scale | 6 weeks
  The total score range of the scale is between 0 and 52. A high total score indicates that the patient's fatigue is low, while a low total score indicates that the patient's fatigue is high. Items 1, 2, 3, 4, 5, 6, 9, 10, 11, 12, and 13 of the scale are reverse scored, while items 7 and 8 are subject to a direct scoring system. The Cronbach's alpha coefficient of the scale was found to be 0.98. In the item analysis results of the scale, all correlations between the items were significantly high. Exploratory factor analysis methods were used to determine the construct validity of the scale, and the factor loading values of all items were found to be between 0.61 and 0.81. According to the factor analysis results, unlike the original scale, two sub-dimensions were found in the Turkish version of the scale. A general score total of less than 30 indicates severe fatigue.
Pittsburg Sleep Quality (PSQI) Scale | 6 weeks
  This scale consists of a total of 24 questions; 19 of these include the individual's own sleep experience, while 5 are answered by the spouse or roommate. Question 19 of the scale does not affect the results. The PSQI includes seven different components that evaluate subjective sleep quality, sleep onset time, sleep duration, sleep efficiency, sleep problems, use of sleeping pills, and daily functioning level. Each component is scored between 0 and 3, and the total score of the scale varies between 0 and 21. (MY, 1996; Roth & Drake, 2004) If the total score of the PSQI is 5 or higher, it reflects poor sleep quality. The Cronbach's Alpha internal consistency coefficient was found to be 0.80. The diagnostic sensitivity of this scale was determined as 89.6% and the specificity as 86.5%.

CONTACTS AND LOCATIONS:
Overall Officials: eren k Kılıç, Principal Investigator — Ataturk University
Locations (1):
- University, Ataturk University Campus, 25030 Yakutiye, Erzurum, Erzurum, Turkey (Türkiye)